CLINICAL TRIAL: NCT00802347
Title: Controlled, Randomized, Prospective, Double-Blind, Multicenter, Phase I/II, Dose-Escalation Study of the Safety, PK, and Clinical Activity of I5NP for Prophylaxis of Delayed Graft Function in Patients Undergoing Deceased Donor Kidney Transplantation
Brief Title: I5NP for Prophylaxis of Delayed Graft Function in Kidney Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Quark Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QRK.006
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Delayed Graft Function; Other Complication of Kidney Transplant
Keywords: Delayed Graft Function; Kidney Transplant; Renal Transplant; small interfering ribonucleic acid (siRNA)
MeSH Terms: conditions — Delayed Graft Function | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I5NP (Experimental)
  Interventions: Drug: I5NP
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: I5NP — Single IV injection of I5NP
  Part A: dose-escalation study; cohort 1 = 0.5 mg/kg; cohort 2 = 1.5 mg/kg; cohort 3 = 5.0 mg/kg; cohort 4 = 10.0 mg/kg
  Part B: 10.0 mg/kg
  Other Names: QPI-1002
  Arms: I5NP
Drug: Saline — Single IV injection of saline
  Part A: dose-escalation study; cohort 1 = 0.5 mg/kg; cohort 2 = 1.5 mg/kg; cohort 3 = 5.0 mg/kg; cohort 4 = 10.0 mg/kg
  Part B: 10.0 mg/kg
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether a single administration of QPI-1002 (also known as I5NP) can prevent DGF in patients undergoing deceased donor kidney transplantation. In this Phase I /II study, patients who are undergoing renal transplantation with organs from DCD donors, ECD donors or SCD donors with ≥ 24 hours of cold ischemia time who meet study entry criteria will be studied to evaluate the safety and pharmacokinetic profile of I5NP (Part A) and clinical activity of I5NP administration (Part B). Data from this study will be used to identify doses of I5NP to be used in follow-on efficacy studies.

Part A will be a randomized, dose escalation study to determine the highest or maximum tolerated dose (MTD). Part A will enroll 40 patients at approximately 20 sites; patients will be randomized to receive either I5NP or placebo in a ratio of 8:2 in each cohort (cohorts 1-4).

Part B will utilize the dose identified in Part A to further evaluate, in a double-blind manner, the safety, and clinical activity of I5NP. In Part B, up to 326 patients will participate at approximately 60 sites; up to 163 patients will be randomized to receive I5NP and up to 163 patients randomized to receive placebo.

DETAILED DESCRIPTION:
Although the etiology of DGF is not fully understood and may be multifactorial, the pathophysiology appears to be primarily related to ischemia-reperfusion (IR) injury resulting from organ preservation between the times of harvesting from the donor and reperfusion following vascular reanastomosis in the recipient.

I5NP is a small interfering RNA (siRNA) that is being developed for the prophylaxis of delayed graft function (DGF) in patients receiving renal transplants.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years of age.
2. Patient has given informed consent.
3. Patient is willing to practice birth control. Female patients must be: (1) post-menopausal (2) surgically sterile, or (3) using an effective means of contraception (per the site-specific guidelines or using 2 methods of birth control concurrently, whichever is more stringent) which will be continued until the Study Day 90 visit with a negative pregnancy test within 48 hours prior to administration of study drug. Male patients with female partners of child bearing potential must agree to use an effective means of contraception (per the site-specific guidelines or using 2 methods of birth control concurrently, whichever is more stringent) which will be continued until the Study Day 90 visit. Note: For the purpose of this study, post menopausal is defined as the absence of menses consistent with ESRD. A woman is considered to be surgically sterilized if she has had a bilateral tubal ligation for at least 6 months prior to administration of study drug, bilateral oophorectomy, or complete hysterectomy.
4. Women of childbearing potential test negative for pregnancy (either urine or serum) within 48 hours prior to transplant.
5. Patient is up-to-date on cancer screening according to site-specific guidelines and the past medical history is negative for biopsy-confirmed malignancy within 5 years of randomization, with the exception of adequately treated basal cell or squamous cell carcinoma in situ.
6. Patient is scheduled to receive kidney transplant from a deceased donor meeting the following criteria:

   Part A:
   * receipt of an extended criteria donor (ECD) kidney, or
   * receipt of a kidney donated after cardiac death (DCD), or
   * receipt of a standard criteria donor (SCD) with cold ischemia time (CIT) ≥ 24 hours.

   Part B:
   * receipt of an ECD kidney that has been preserved by cold storage (ECD/CS) for the entire period of cold ischemia time (CIT), regardless of duration
   * receipt of an ECD kidney that has been preserved by machine perfusion (ECD/MP) for any interval of time during the period of cold ischemia, where total CIT has been at least 26 hours
   * receipt of an SCD kidney that has been preserved by cold storage (SCD/CS) where total CIT has been at least 26 hours
   * receipt of an SCD kidney that has been preserved by machine perfusion (SCD/MP) for any interval of time during the period of cold ischemia, where total CIT has been at least 26 hours.
7. Patient is dialysis dependent at the time of transplant as documented by: a) the requirement for at least 2 dialysis sessions/week during the 56 days prior to transplant, or b) the planned removal of any remaining native kidney at the time of transplant, or c) the opinion of the investigator that the patient has no remaining native renal function (Part A only), or d) the investigator has provided documentation to the Medical Monitor that the patient has no remaining native renal function (e.g., documentation that the patient is anuric, with urine output <50 mL/day) (Part B only).

Exclusion Criteria:

1. Patient has participated in an investigational drug study in the last 30 days.
2. Patient has known allergy or has participated in prior study with siRNA.
3. Patient is HCV-positive
4. Patient is HIV-positive
5. Patient is scheduled to undergo multiorgan transplantation.
6. Patient has a planned transplant of kidneys that are implanted en bloc (dual kidney transplant).
7. Patient has planned transplant of kidneys from donors < 6 years of age.
8. Patient has planned transplant of dual kidneys (from the same donor) transplanted not en bloc (as in the case of dual ECD donor kidneys).
9. Patient is scheduled for transplantation of a kidney from a donor who is known to have received an investigational therapy (under another IND) for ischemic/reperfusion injury immediately prior to organ recovery.
10. Patient is scheduled to receive a living donor kidney.
11. Patient is scheduled to receive an ABO-incompatible donor kidney.
12. Patient is scheduled to receive an organ from a donor that meets both DCD and ECD criteria.
13. Patient is scheduled to receive an organ from a donor that meets DCD criteria (exclusion applicable to Part B only).
14. Patient has history or presence of a medical condition or disease that in the investigator's assessment would place the patient at an unacceptable risk for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2008-12; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Part A: The outcome measure is safety. Additionally, plasma blood levels will be measured to characterize the PK of I5NP in this patient population. Part B: The outcome measure will be safety and the incidence of delayed graft function. | Part A: DSMB review at conclusion of each cohort / Part B: Interim analyses will be performed after the 66th, 130th, and 196th patient enrolled

SECONDARY OUTCOMES:
Part B: Treatment differences in the rate of improvement in renal function over time and treatment differences in the need for renal replacement therapy. | Part B: Interim analyses will be performed after the 66th, 130th, and 196th patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Shai Erlich, Ph.D., Study Director — Quark Pharmaceuticals
Locations (50):
- United States (33):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Transplant Research Institute (TRI; formerly NIT), Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - University of Colorado Health Science Center, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Lifelink Healthcare Institute, Tampa, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - University of Illinois Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Columbia University, New York, New York
  - Cornell University, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University Medical Center, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University (MCV), Richmond, Virginia
- Canada (4):
  - St. Paul's Hospital, Univeristy of BC, Vancouver, British Columbia
  - UBC - Division of Nephrology, Vancouver, British Columbia
  - QE II Capital District Health Authority, Halifax, Halifax, Nova Scotia
  - MUHC Royal Victoria Hospital, Montreal, Quebec
- France (3):
  - Hôpital Pasteur, Nice
  - Hôpital Necker, Paris
  - CHU Rangueil, Toulouse
- Germany (7):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Charité, Campus Virchow-Klinikum, Berlin
  - Kliniken der Stadt Köln gGmbH, Cologne
  - Universitätklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Tübingen, Tübingen
- Spain (3):
  - Hospital de bellvitge, Barcelona
  - Hospital del mar, Barcelona
  - Hospital Vall Hebron, Barcelona